CLINICAL TRIAL: NCT05407155
Title: BEvacizumab Plus Nab-pacliTaxel and plaTinum as sEcond-line theRapy for Driver-gene-negative Non-squamous Non-small Cell Lung Cancer Progressed After First-line Immune Checkpoint Inhibitor-based Regimen
Brief Title: Bevacizumab Plus Nab-paclitaxel and Platinum for Immunotherapy-treated Non-squamous Non-small Cell Lung Cancer
Acronym: BETTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Associate Director of Department of Thoracic Medical Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BETTER-NSCLC-2021
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Bevacizumab; 130-nm albumin-bound paclitaxel; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients received bevacizumab plus nab-paclitaxel and platinum as second-line therapy.
  Interventions: Combination Product: bevacizumab plus nab-paclitaxel and platinum

INTERVENTIONS:
Combination Product: bevacizumab plus nab-paclitaxel and platinum — Bevacizumab is given as 15mg/kg every 3 weeks. Nab-paclitaxel is given as 260 mg/m2 every 3 weeks for 4 cycles at most. Platinum includes caboplatin or cisplatin, which is chosed by phycisians. Carboplatin was calculated using AUC equals 5 for 4 cycles at most, and cisplatin was given as 75mg/m2 for 4 cycles at most. Bevacizumab is given untill disease progression or intolerated toxicities.

SUMMARY:
Immune checkpoint inhibitor (ICI)-based regimen has been widely used in first-line treatment of driver-gene-negative non-squamous non-small cell lung cancer. This study investigate the efficacy and safety of the combination of bevacizumab plus nab-paclitaxel and platinum as second-line treatment for driver-gene-negative non-squamous non-small cell lung cancer patients progressed after ICI-based treatments.

ELIGIBILITY:
Inclusion Criteria:

1. The participants voluntarily signed the informed consent form.
2. The participants should be 18~75 years old.
3. Histology or cytology confirmed, stage IIIB to IV non-small cell lung cancer (according to the eighth edition of the American Joint Committee on cancer AJCC staging) that could not undergo radical treatment.
4. No sensitive EGFR mutation, ALK gene rearrangement and ROS1 gene rearrangement are allowed.
5. Progressed after first-line treatment included immune checkpoint inhibitor (including CTLA-4 monoclonal antibody, PD-1/L1 monoclonal antibody monothrapy or combination therapy, with or without chemotherapy. If the first-line treatment is discontinued due to adverse effects, and patients received no other treatment before disease progression.
6. For patients who have previously received neoadjuvant and/or adjuvant immune checkpoint inhibitor treatment (with or without chemotherapy or radiotherapy) for the purpose of radical treatment of non-metastatic disease, if first-line treatment contained immune checkpoint inhibitors (the same or different immune checkpoint inhibitors with neoadjuvant or adjuvant settings), they can also be included.
7. At least one measurable lesion according to RECIST criteria v1.1. If patients received radiotherapy, they can be included only when disease progression of the previously irradiated lesion is observed, and the previously irradiated lesion is not the only lesions.
8. ECOG PS score: 0-1.
9. The estimated survival time is more than 3 months.
10. Laboratory test results showed sufficient hematology and end organ functions.
11. Patients with asymptomatic central nervous system (CNS) metastases can be enrolled. Patients with symptomatic CNS metastases should received local treatment and meet the following conditions before enrollment: a) stable for at least 14 days before enrollment with or without receiving steroids and anticonvulsant drugs; b) Complete radiotherapy at least 14 days before enrollment; c) From the end of radiotherapy to the screening phase, no CNS progression was found. If local CNS treatment is performed before enrollment, there should be at least one extracranial measurable lesion according to RECIST criteria v1.1.
12. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; Within 7 days before the study, the serum or urine pregnancy test was negative; Non-lactating patients; Men should agree to use contraceptives during the study period and within 6 months after the end of the study period.
13. Ability to follow research and follow-up procedures.

Exclusion Criteria:

1. Histologically mixed with small cell or squamous lung cancer.
2. Previously received anti-angiogenic drugs (including bevacizumab, arotinib, apatinib, etc.) and/or paclitaxel (including paclitaxel, paclitaxel liposomes, and nab-paclitaxel). If paclitaxel is used in the adjuvant treatment setting, patients who progressed after 6 months from the last dose of paclitaxel can be included.
3. Patients diagnosed with secondary primary malignant tumor within 5 years before enrollment, except cured cervical carcinoma in situ, superficial bladder tumor [Ta, Tis and T1], basal or squamous cell skin cancer, localized prostate cancer after radical surgery and breast ductal carcinoma in situ after radical surgery.
4. Patients with leptomeningeal metastasis or untreated symptomatic or rapidly progressing CNS metastasis.
5. Unrelieved toxic reactions of CTCAE (5.0) grade 2 or higher caused by any previous treatments, excluding hair loss, nausea and vomiting.
6. For uncontrollable tumor-related pain, patients who need analgesic treatment must have a stable analgesic treatment plan at enrollment. If there are symptomatic lesions suitable for palliative radiotherapy (such as bone metastasis or metastatic nerve invasion), the treatment should be completed before enrollment. The patient should recover from the effects of radiation. For asymptomatic metastatic lesions, if the investigator believes there is the possibility of dysfunction or intractable pain (such as epidural metastasis not currently related to spinal cord compression), local regional treatment should be considered before enrollment.
7. Major surgery other than that for the purpose of diagnosis was performed within 4 weeks before enrollment, or expected major surgery during the study period.
8. Serious infection within 4 weeks before enrollment, including but not limited to infection, bacteremia or severe pneumonia that leads to hospitalization, or any active infection that the investigator believes may affect the safety of patients.
9. Patients with any severe and / or uncontrolled disease, including:

(1) Patients with unsatisfactory blood pressure control (systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg), hypertensive crisis or hypertensive encephalopathy; (2) Major cardiovascular diseases, including but not limited to: myocardial ischemia or myocardial infarction above grade I, arrhythmia (including QTc ≥ 440ms) and congestive heart failure ≥ grade 2 (NYHA classification); (3) Active or uncontrolled severe infection (≥ CTCAE grade 2 infection); (4) Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation; (5) Uncontrolled pleural effusion, pericardial effusion and peritoneal effusion requiring repeated drainage (once a month or more frequently); (6) Poor control of diabetes [fasting blood glucose (FBG) > 10mmol/l]; (7) Urine routine examination showed that urine protein was ≥++, and the 24-hour urine protein was confirmed to be more than 1.0 G; (8) Patients who have seizures and need treatment; (9) Uncontrolled or symptomatic hypercalcemia (ionic calcium > 1.5 mmol/l, calcium > 12 mg/dl or corrected serum calcium > ULN).

10. Arteriovenous thrombosis events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism within 6 months before enrollment.

11. Hemoptysis ≥ grade 2 (defined as ≥ 2.5 ml of bright red blood each time) within 3 months before enrollment.

12. Bleeding tendencies or coagulation disorders (i.e. without the use of therapeutic anticoagulants).

13. Tumor infiltration or adjacency to large blood vessels. 14. A history of abdominal fistula, gastrointestinal (GI) perforation, abdominal abscess, or active gastrointestinal bleeding within 6 months before enrollment.

15. Aspirin (> 325 mg/d) or clopidogrel (> 75 mg/d) was used currently or recently (10 days before starting the study treatment). The preventive use of anticoagulants is permitted.

16. Active pulmonary tuberculosis (TB) or subjects with a history of active TB infection within ≤ 48 weeks before enrollment, whether treated or not.

17. Have a history of idiopathic pulmonary fibrosis, organized pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, radiation pneumonia requiring steroid treatment or active pneumonia with clinical symptoms; Or other moderate or severe lung diseases that seriously affect lung function.

18. Has a history of psychotropic substance abuse and is unable to quit or has mental disorders.

19. Known history of allergic or hypersensitive to any component of carboplatin / cisplatin or bevacizumab, and there are no other alternative drugs allowed by this protocol. Patients who are known to be allergic to paclitaxel can be enrolled if clinicians decide that nab-paclitaxel could be used.

20. Pregnant or lactating women. 21. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From enrollment to end of study, up to 2 years
  Proportion of patients achieved complete response or partial response

SECONDARY OUTCOMES:
Progression free survival | From enrollment to date of disease progression or death of any cause, regardless of whichever would occur first, up to 2 years
  The time duration of patients from enrollment to date of disease progression or death of any cause, regardless of whichever would occur first.
Overall survival | From enrollment to date of death of any cause, up to 2 years
  The time duration of patients from enrollment to date of death of any cause.

IPD SHARING:
Plan to Share IPD: No